CLINICAL TRIAL: NCT03288896
Title: Alerta Alcohol. Design, Implementation, and Evaluation of a Tailored Web-based Computer-tailored Intervention for Selective Prevention of Binge-drinking in Spanish Adolescents.
Brief Title: Alerta Alcohol. Web-based Computer-tailored Intervention for Binge-drinking Prevention in Spanish Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Junta de Andalucia (Other Government); Maastricht University (Other)
Responsible Party: Principal Investigator, Marta Lima Serrano, PhD, University of Seville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: University of Seville. Spain
Record Dates: First submitted 2017-09-17; First posted 2017-09-20 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Alcohol Drinking; Binge Drinking; Adolescent Behavior
Keywords: Adolescence; Alcohol Drinking; Binge Drinking; I-Change model; Web-based interventions; Computer-tailoring
MeSH Terms: conditions — Alcohol Drinking; Binge Drinking; Adolescent Behavior | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: A Cluster Randomized Controlled Trial is conducted to test the effectiveness of Alerta Alcohol in students aged 16 to 18 years. The study is performed in 16 high schools from Andalusia (southern Spain), which are randomized either to the experimental or the control condition (EC and CC). The EC receives the Alerta Alcohol intervention, which consists of four sessions at school. The adolescents are provided highly specific feedback regarding their knowledge, risk perception, self-esteem, attitude, social influence, and self-efficacy. In addition, two booster sessions are given at home to reinforce the contents of the three scenarios. The CC just completes the baseline and the evaluation questionnaires and then they are allowed to receive the intervention as well (as a waiting list control condition).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alerta Alcohol (Experimental): Intervention Group: The Experimental Group receives the Alerta Alcohol intervention, which consists of four sessions at school (baseline questionnaire, two sessions in three scenarios: at home, celebrations, and public places, and a final evaluation). The adolescents are provided with answers related to their views of each scenario; this information is used to provide highly specific feedback regarding their knowledge, risk perception, self-esteem, attitude, social influence (modelling, norms and social pressure), self-efficacy and action plans. In addition, two booster sessions are given at home to reinforce the contents of the three scenarios. Evaluation takes place after four months.
  Interventions: Behavioral: Alerta Alcohol
- Control Group (No Intervention): Control Group: The Control Group just completes the baseline and the evaluation questionnaires and then they are allowed to receive the intervention as well (as a waiting list control condition). Evaluation takes place after four months from baseline

INTERVENTIONS:
Behavioral: Alerta Alcohol — The intervention consists of preventive messages about the benefits of not consuming alcohol, reducing the positive attitudes and encouraging the negative attitudes towards alcohol drinking and binge drinking, as well as social influence and self-efficacy, by personalized feedback. Skills and action plans are encouraged to help the student to reject binge drinking. This information is presented through different tailored messages. Moreover, four avatars (two males and two females), which can be chosen as part of the story development. This story consists of a short story about the alcohol consumption by adolescents.The stories take place in three different scenarios (at home, at celebrations and in public places).
  Other Names: Alerta Alcohol, a web-based computer-tailored intervention
  Arms: Alerta Alcohol

SUMMARY:
This study consists in the the design, implementation, and evaluation of the first web-based computer tailored intervention program aimed at the prevention of binge drinking in Spanish adolescents (Alerta Alcohol). A Cluster Randomized Controlled Trial is conducted to test the effectiveness of Alerta Alcohol in students aged 16 to 18 years across 16 high schools from Andalusia (southern Spain), which are randomized either to the experimental or the control condition (EC and CC).

DETAILED DESCRIPTION:
Binge-drinking in adolescents is a highly prevalent healthcare problem that associates physical and mental health complications and community implications.

The "Alerta Alcohol" program is based on the I-Change Model. Focus and Delphi groups are used to obtain further information on items included in the program. A pilot study is conducted to identify strengths and weaknesses. A Cluster Randomized Controlled Trial is carried out. The schools from Andalusia are randomized either to the experimental or the control condition (EC and CC). The EC receives the Alerta Alcohol intervention, which consists of four sessions at school: baseline questionnaire and two sessions where adolescents are provided with answers related to their views to provide highly specific feedback regarding their knowledge, risk perception, self-esteem, attitude, social influence, and self-efficacy. In addition, two booster sessions are given at home to reinforce the contents. The CC just completes the baseline and the evaluation questionnaires and then they are allowed to receive the intervention as well (as a waiting list control condition). Evaluation takes place after four months. The primary endpoint is binge drinking within 30 days prior to evaluation and alcohol use in the previous week. It is expected that Alerta Alcohol reduces the prevalence of binge drinking by 10%. Follow up analyses are carried out to determine the differences in effectiveness according to the compliance of the program (quality of the implementation).

ELIGIBILITY:
Inclusion Criteria:

* Students aged 16 to 18 years.
* Enrolled in Andalusian public high schools.
* Schools belonging to provincial capitals.
* Access to the Internet at the school and an equipped ICT room.

Exclusion Criteria:

* Language barriers.
* Previous participation in prevention programs for binge drinking.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1230 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Reducing binge-drinking | 4 months after the baseline
  Reducing binge-drinking (4/5 glasses or alcohol in one ocassion for a girl/boy) within 30 days prior to evaluation.

SECONDARY OUTCOMES:
Reducing weekly alcohol drinking | 4 months after the baseline
  Reducing alcohol drinking within the 7 days prior to evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Marta Lima Serrano, PhD, Study Director — University of Seville
Locations (1):
- Marta Lima Serrano, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared with other researchers through publications in scientific journals and congresses
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From 2018
Access Criteria: The Access Criteria will be the one exposed by the scientific journals where the results of the study will be published.

REFERENCES:
- [Derived] Vargas-Martinez AM, Lima-Serrano M, Trapero-Bertran M. Cost-effectiveness and cost-utility analyses of a web-based computer-tailored intervention for prevention of binge drinking among Spanish adolescents. Alcohol Clin Exp Res (Hoboken). 2023 Feb;47(2):319-335. doi: 10.1111/acer.14990. Epub 2023 Feb 22. PMID 36811462
- [Derived] Vargas-Martinez AM, Trapero-Bertran M, Mora T, Lima-Serrano M. Social, economic and family factors associated with binge drinking in Spanish adolescents. BMC Public Health. 2020 Apr 17;20(1):519. doi: 10.1186/s12889-020-08605-9. PMID 32303203
- [Derived] Martinez-Montilla JM, Mercken L, de Vries H, Candel M, Lima-Rodriguez JS, Lima-Serrano M. A Web-Based, Computer-Tailored Intervention to Reduce Alcohol Consumption and Binge Drinking Among Spanish Adolescents: Cluster Randomized Controlled Trial. J Med Internet Res. 2020 Jan 24;22(1):e15438. doi: 10.2196/15438. PMID 32012064
- [Derived] Vargas-Martinez AM, Trapero-Bertran M, Lima-Serrano M, Anokye N, Pokhrel S, Mora T. Measuring the effects on quality of life and alcohol consumption of a program to reduce binge drinking in Spanish adolescents. Drug Alcohol Depend. 2019 Dec 1;205:107597. doi: 10.1016/j.drugalcdep.2019.107597. Epub 2019 Sep 30. PMID 31590139
- [Derived] Lima-Serrano M, Martinez-Montilla JM, Lima-Rodriguez JS, Mercken L, de Vries H. Design, implementation and evaluation of a web-based computer-tailored intervention to prevent binge drinking in adolescents: study protocol. BMC Public Health. 2018 Apr 4;18(1):449. doi: 10.1186/s12889-018-5346-4. PMID 29618331